CLINICAL TRIAL: NCT01945216
Title: Alogliptin Tablets Special Drug Use Surveillance "Type 2 Diabetes Mellitus: Monotherapy/Combination Therapy With α-GI"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 121-011; JapicCTI-132250 (Registry Identifier: JapicCTI); JapicCTI-R171018 (Other: JapicCTI)
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Type 2 Diabetes Mellitus Who Have Been Examined at a Medical Institution
Keywords: Drug therapy
MeSH Terms: interventions — alogliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alogliptin 25mg, tablets, orally, once daily, up to 36 months
  Interventions: Drug: Alogliptin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: Nesina; SYR-322

SUMMARY:
The purpose of this study is to determine the safety and efficacy of long-term treatment with alogliptin (Nesina) in patients with type 2 diabetes mellitus who responded inadequately to diet therapy and exercise therapy alone, or a combination of diet therapy, exercise therapy, and α-glucosidase inhibitor.

In addition, examining the safety and efficacy of alogliptin in patients with renal impairment, information on the appropriate dosage of alogliptin according to the severity of impaired renal function should be collected.

DETAILED DESCRIPTION:
A special drug use surveillance is planned to examine the safety and efficacy of long-term use of alogliptin in patients with type 2 diabetes mellitus under the daily clinical use conditions.

Participants of this surveillance will be patients with type 2 diabetes mellitus who failed to respond adequately to diet therapy and exercise therapy alone or to a combination of diet therapy, exercise therapy, and α-glucosidase inhibitor. The planned sample size is 3,000 subjects.

The usual adult dosage for oral use is 1 alogliptin tablet (25 mg) once daily. Participants will receive the drug as part of routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus who have not adequately responded to any one of the following therapies:

  1. Diet therapy and exercise therapy alone
  2. In addition to diet therapy and exercise therapy, use of α-glucosidase inhibitor

Exclusion Criteria:

* Patients contraindicated for Nesina

  1. Patients with severe ketosis, diabetic coma or precoma, or type 1 diabetes mellitus (these patients require prompt adjustment of hyperglycemia by fluid infusion and insulin, and hence use of Nesina is not appropriate.)
  2. Patients with severe infection, pre- or post-operative patients, or patients with serious traumatic injury (blood glucose control by insulin injection is desirable for these patients, and hence use of Nesina is not appropriate.)
  3. Patients with a history of hypersensitivity to any ingredient of Nesina

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus who have been examined at a medical institution
Sampling Method: Non-Probability Sample
Enrollment: 3317 (Actual)
Dates: Start 2010-07-08 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Osaka, Japan

IPD SHARING:
Plan to Share IPD: No
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 608 investigative sites in Japan, from 8-July-2010 to 31-October-2015. Data reports overall population, since data not collected separately per arm as specified in protocol.
Pre-assignment Details: Participants with type 2 diabetes mellitus who failed to respond adequately to diet and/or exercise therapy and α-glucosidase inhibitor were enrolled to receive Alogliptin as routine medical care. Treatments were not allocated at the start of the study. Thus, the Participant Flow cannot be presented "per Arm".
Groups:
- Overall Population: Alogliptin 25 milligram (mg), tablets, orally, once daily, up to 36 months along with an alpha-glucosidase inhibitor (α-GI), without an α-GI, or the other diabetic drugs from the start of administration of alogliptin and during the treatment period of alogliptin in routine medical care.
Period: Overall Study
Arm/Group | Overall Population
Started | 3317
Completed | 3218
Not Completed | 99
Not completed — Case report forms (CRF) uncollected | 52
Not completed — Protocol Violation | 42
Not completed — CRF not assured by investigators | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Groups:
- Alogliptin: Alogliptin 25 mg, tablets, orally, once daily for up to 36 months in routine medical care. Participants in this group received no diabetic drugs within 3 months from the start of administration of alogliptin and during the treatment period of alogliptin.
- Alogliptin + αGI: Alogliptin 25 mg, tablets, orally, once daily for up to 36 months in routine medical care. Participants in this group received an α-GI within 3 months from the start of administration of alogliptin and during the treatment period of alogliptin.
- Alogliptin + Other: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months in routine medical care. Participants in this group did not receive an α-GI within 3 months from the start of administration of alogliptin or during the treatment period of alogliptin.
- Total: Total of all reporting groups
Arm/Group | Alogliptin | Alogliptin + αGI | Alogliptin + Other | Total
Number analyzed (Participants) | 1560 | 669 | 989 | 3218
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (12.28) | 67.1 (12.13) | 64.0 (12.57) | 65.1 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 640 | 286 | 438 | 1364
  Male | 920 | 383 | 551 | 1854
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 1560 | 669 | 989 | 3218
Time From Diagnosis of Type 2 Diabetes [Mean (Standard Deviation); unit: years] — Population: The number analyzed is the number of participants with data available for analysis.
  years
    number analyzed (Participants) | 1161 | 501 | 722 | 2384
    (all) | 3.45 (4.923) | 8.10 (7.018) | 5.03 (5.732) | 4.91 (5.937)
Height [Mean (Standard Deviation); unit: cm] — Population: The number analyzed is the number of participants with data available for analysis.
  cm
    number analyzed (Participants) | 1439 | 621 | 894 | 2954
    (all) | 160.22 (9.686) | 159.33 (9.535) | 160.18 (9.738) | 160.02 (9.674)
Body Weight [Mean (Standard Deviation); unit: kg] — Population: The number analyzed is the number of participants with data available for analysis.
  kg
    number analyzed (Participants) | 1538 | 664 | 976 | 3178
    (all) | 64.49 (13.699) | 62.68 (13.005) | 64.51 (14.046) | 64.12 (13.681)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  kg/m^2
    number analyzed (Participants) | 1431 | 619 | 889 | 2939
    (all) | 25.00 (4.225) | 24.52 (4.277) | 25.04 (4.190) | 24.91 (4.229)
Waist Circumference (Male) [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in male participants.
  Participants
    number analyzed (Participants) | 920 | 383 | 551 | 1854
    < 85cm | 96 | 55 | 61 | 212
    ≥ 85cm | 211 | 80 | 120 | 411
    Unknown | 613 | 248 | 370 | 1231
Waist Circumference (Female) [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    number analyzed (Participants) | 640 | 286 | 438 | 1364
    < 90cm | 152 | 65 | 85 | 302
    ≥ 90cm | 70 | 37 | 52 | 159
    Unknown | 418 | 184 | 301 | 903
Healthcare category [Count of Participants; unit: Participants] — Participants were categorized as outpatient, inpatient, and In- to/from out-patient (participants who were both outpatient and inpatient at any time prior to enrollment).
  Participants
    Out-patient | 1524 | 640 | 942 | 3106
    In-patient | 3 | 8 | 11 | 22
    In- to/from out-patient | 33 | 21 | 36 | 90
Pregnancy Status [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    number analyzed (Participants) | 640 | 286 | 438 | 1364
    Not pregnant | 640 | 286 | 438 | 1364
    Pregnant | 0 | 0 | 0 | 0
History of Allergy [Count of Participants; unit: Participants]
  Had no history of Allergy | 1377 | 583 | 856 | 2816
  Had history of Allergy | 127 | 57 | 104 | 288
  Unknown | 56 | 29 | 29 | 114
Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Complications | 314 | 61 | 103 | 478
    Had Complications | 1246 | 608 | 886 | 2740
Diabetic Complications [Count of Participants; unit: Participants]
  Had No Diabetic Complications | 1402 | 506 | 831 | 2739
  Had Diabetic Complications | 158 | 163 | 158 | 479
Hypertension Complications [Count of Participants; unit: Participants]
  Had No Hypertension Complications | 676 | 249 | 383 | 1308
  Had Hypertension Complications | 884 | 420 | 606 | 1910
Hyperlipidemia Complications [Count of Participants; unit: Participants]
  Had No Hyperlipidemia Complications | 715 | 246 | 375 | 1336
  Had Hyperlipidemia Complications | 845 | 423 | 614 | 1882
Hyperuricemia Complications [Count of Participants; unit: Participants]
  Had No Hyperuricemia Complications | 1411 | 611 | 891 | 2913
  Had Hyperuricemia Complications | 149 | 58 | 98 | 305
Hepatic Dysfunction Complications [Count of Participants; unit: Participants]
  Had No Hepatic Dysfunction Complications | 1322 | 553 | 799 | 2674
  Had Hepatic Dysfunction Complications | 238 | 116 | 190 | 544
Degree of Hepatic Dysfunction [Count of Participants; unit: Participants] — Severity was determined using aspartate aminotransferase (AST) or alanine transaminase (ALT) values at the start of treatment with alogliptin. For the assessment of severity, the following categories were used and higher grades of serum AST or ALT were adopted. Normal: <50 international units per liter (IU/L) Grade 1: >=50 to <100 IU/L Grade 2: >=100 to <500 IU/L Grade 3: >=500 IU/L
  Participants
    Normal | 986 | 443 | 596 | 2025
    Grade 1 | 122 | 36 | 87 | 245
    Grade 2 | 22 | 10 | 19 | 51
    Grade 3 | 0 | 0 | 0 | 0
    Unknown | 430 | 180 | 287 | 897
Renal Dysfunction Complications [Count of Participants; unit: Participants]
  Had No Renal Dysfunction Complications | 1427 | 563 | 861 | 2851
  Had Renal Dysfunction Complications | 133 | 106 | 128 | 367
Degree of Renal Dysfunction (eGFR) [Count of Participants; unit: Participants] — Estimated glomerular filtration rate (eGFR) was calculated using variables of gender, age at the start of treatment, and serum creatinine values, and severity was determined based on the following categories. If the serum creatinine value at the start of treatment was not listed, the severity was reported as "unknown." Normal: >=90 milliliter per min (mL/min)/1.73^2, Mild: >=60 mL/min/1.73^2 to <90 mL/min/1.73^2, Moderate: >=30 mL/min/1.73^2 to <60 mL/min/1.73^2, Severe: <30 mL/min/1.73^2 eGFR = 194 * Cr^-1.094 * (age)^-0.287 (* 0.739 if female) where Cr is creatinine value.
  Participants
    Normal | 249 | 108 | 189 | 546
    Mild | 667 | 254 | 361 | 1282
    Moderate | 190 | 108 | 121 | 419
    Severe | 28 | 22 | 25 | 75
    Unknown | 426 | 177 | 293 | 896
Degree of Renal Dysfunction (Cr) [Count of Participants; unit: Participants] — Normal or Mild: =< 1.4 mg/dL (for male) or =< 1.2 mg/dL (for female), Moderate: >1.4 mg/dL to =< 2.4 mg/dL (for male) or >1.2 mg/dL to =< 2.0 mg/dL (for female), Severe: > 2.4 mg/dL (for male), > 2.0 mg/dL (for female). If the serum creatinine value (Cr) at the start of treatment was not listed, the severity was reported as "unknown."
  Participants
    Normal or Mild | 1089 | 466 | 664 | 2219
    Moderate | 24 | 7 | 17 | 48
    Severe | 21 | 19 | 15 | 55
    Unknown | 426 | 177 | 293 | 896
Cardiac Disease Complications [Count of Participants; unit: Participants]
  Had No Cardiac Disease Complications | 1417 | 578 | 870 | 2865
  Had Cardiac Disease Complications | 143 | 91 | 119 | 353
Heart Failure Complications [Count of Participants; unit: Participants]
  Had No Heart Failure Complications | 1517 | 649 | 970 | 3136
  Had Heart Failure Complications | 43 | 20 | 19 | 82
New York Heart Association (NYHA) Heart Failure Classification [Count of Participants; unit: Participants] — NYHA functional classification ranges from Class I (Participants with cardiac disease but without resulting limitations of physical activity), Class II (Participants with cardiac disease resulting in slight limitation of physical activity), Class III (Participants with cardiac disease resulting in marked limitation of physical activity), Class IV (Participants with cardiac disease resulting in inability to carry on any physical activity without discomfort). Population: This baseline characteristic was analyzed only for Participants who had complications of heart failure.
  Participants
    number analyzed (Participants) | 43 | 20 | 19 | 82
    NYHA Class I | 26 | 13 | 11 | 50
    NYHA Class II | 16 | 5 | 5 | 26
    NYHA Class III | 1 | 1 | 1 | 3
    NYHA Class IV | 0 | 0 | 0 | 0
    Unknown | 0 | 1 | 2 | 3
Stroke-Related Disorder Complications [Count of Participants; unit: Participants]
  Had No Stroke-Related Disorder Complications | 1505 | 613 | 922 | 3040
  Had Stroke-Related Disorder Complications | 55 | 56 | 67 | 178
Allergic Disease Complications [Count of Participants; unit: Participants]
  Had No Allergic Disease Complications | 1466 | 627 | 914 | 3007
  Had Allergic Disease Complications | 94 | 42 | 75 | 211
Malignancy Complications [Count of Participants; unit: Participants]
  Had No Malignancy Complications | 1543 | 661 | 960 | 3164
  Had Malignancy Complications | 17 | 8 | 29 | 54
Medical history [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had No Medical History | 1255 | 501 | 768 | 2524
    Had Medical History | 225 | 126 | 166 | 517
    Unknown | 80 | 42 | 55 | 177
Alcohol Consumption Classification [Count of Participants; unit: Participants]
  Drinking Almost Everyday | 412 | 158 | 276 | 846
  Not Drinking Almost Everyday | 891 | 383 | 526 | 1800
  Unknown | 257 | 128 | 187 | 572
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 737 | 292 | 414 | 1443
  Current Smoker | 227 | 77 | 155 | 459
  Ex-Smoker | 249 | 153 | 160 | 562
  Unknown | 347 | 147 | 260 | 754
Glycosylated Hemoglobin A1c (HbA1c) [Count of Participants; unit: Participants]
  HbA1c <6.0 percent | 28 | 24 | 33 | 85
  HbA1c >=6.0 to <7.0 percent | 475 | 134 | 195 | 804
  HbA1c >=7.0 to <8.0 percent | 576 | 270 | 320 | 1166
  HbA1c >=8.0 percent | 351 | 195 | 345 | 891
  Unknown | 130 | 46 | 96 | 272

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Adverse Events
Time Frame: Up to Month 36
Population: Safety Analysis Set was defined as all participants who were enrolled and completed the study.
Measure: Count of Participants; unit: Participants
Groups:
- Alogliptin + α-GI: Alogliptin 25 mg, tablets, orally, once daily for up to 36 months in routine medical care. Participants in this group received an α-GI within 3 months from the start of administration of alogliptin and during the treatment period of alogliptin.
Arm/Group | Alogliptin | Alogliptin + α-GI | Alogliptin + Other
Number analyzed (Participants) | 1560 | 669 | 989
Participants | 151 | 98 | 139

2. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at month 36 relative to baseline.
Time Frame: Baseline, Months 1, 3, 6, 12, 18, 24, 30, 36 and final assessment (up to Month 36)
Population: The efficacy assessment population was defined as participants who completed the study and had available efficacy data at baseline and post baseline. Reported group were Alogliptin and Alogliptin + α-GI and data for Alogliptin + Other were not collected as specified in protocol.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Alogliptin | Alogliptin + α-GI
Number analyzed (Participants) | 1341 | 612
Percent
  Change at Month 1: number analyzed (Participants) | 1015 | 504
  Change at Month 1 | -0.45 (0.581) | -0.33 (0.708)
  Change at Month 3: number analyzed (Participants) | 1104 | 535
  Change at Month 3 | -0.79 (1.007) | -0.54 (1.074)
  Change at Month 6: number analyzed (Participants) | 1043 | 526
  Change at Month 6 | -0.84 (1.045) | -0.70 (1.128)
  Change at Month 12: number analyzed (Participants) | 1030 | 498
  Change at Month 12 | -0.83 (1.102) | -0.75 (1.054)
  Change at Month 18: number analyzed (Participants) | 805 | 423
  Change at Month 18 | -0.81 (1.077) | -0.62 (1.190)
  Change at Month 24: number analyzed (Participants) | 753 | 394
  Change at Month 24 | -0.82 (1.095) | -0.66 (1.214)
  Change at Month 30: number analyzed (Participants) | 664 | 353
  Change at Month 30 | -0.83 (1.114) | -0.73 (1.271)
  Change at Month 36: number analyzed (Participants) | 663 | 331
  Change at Month 36 | -0.84 (1.131) | -0.72 (1.318)
  Change at Final Assessment | -0.81 (1.140) | -0.63 (1.381)

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: The change in the value of fasting blood glucose collected at month 36 relative to baseline.
Time Frame: Baseline, Months 1, 3, 6, 12, 18, 24, 30, 36 and final assessment (up to Month 36)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin | Alogliptin + α-GI
Number analyzed (Participants) | 510 | 229
mg/dL
  Change at Month 1: number analyzed (Participants) | 311 | 152
  Change at Month 1 | -22.9 (45.05) | -4.9 (41.17)
  Change at Month 3: number analyzed (Participants) | 358 | 175
  Change at Month 3 | -21.7 (39.40) | -8.3 (36.58)
  Change at Month 6: number analyzed (Participants) | 322 | 171
  Change at Month 6 | -19.1 (36.46) | -14.5 (49.90)
  Change at Month 12: number analyzed (Participants) | 324 | 163
  Change at Month 12 | -23.1 (43.60) | -18.4 (41.37)
  Change at Month 18: number analyzed (Participants) | 234 | 126
  Change at Month 18 | -21.1 (41.54) | -16.0 (46.75)
  Change at Month 24: number analyzed (Participants) | 214 | 119
  Change at Month 24 | -19.9 (42.56) | -14.0 (42.09)
  Change at Month 30: number analyzed (Participants) | 183 | 102
  Change at Month 30 | -24.4 (39.14) | -11.7 (52.27)
  Change at Month 36: number analyzed (Participants) | 201 | 99
  Change at Month 36 | -23.0 (45.19) | -18.6 (48.80)
  Change at Final Assessment | -24.5 (48.45) | -12.2 (51.25)

ADVERSE EVENTS:
Time Frame: Up to Month 36
Description: Reported data on Serious Adverse Events were serious adverse drug reactions since only serious adverse drug reactions were collected in this study as specified protocol. Participants may be represented in more than 1 category.
Arm/Group | Alogliptin | Alogliptin + αGI | Alogliptin + Other
All-Cause Mortality (participants affected / at risk) | 1/1560 | 1/669 | 2/989
Serious Adverse Events (participants affected / at risk) | 2/1560 | 2/669 | 8/989
Other Adverse Events (participants affected / at risk) | 26/1560 | 19/669 | 23/989
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin (N=1560) | Alogliptin + αGI (N=669) | Alogliptin + Other (N=989)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Sudden death (General disorders) | 1 | 0 | 0 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin (N=1560) | Alogliptin + αGI (N=669) | Alogliptin + Other (N=989)
Hypertension (Vascular disorders) | 20 | 13 | 17
Hepatic function abnormal (Hepatobiliary disorders) | 6 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.